CLINICAL TRIAL: NCT06213311
Title: A Phase 2 Study of Axicabtagene Ciloleucel and Glofitamab as Second-Line Therapy for Relapsed or Refractory Patients With Large B Cell Lymphoma
Brief Title: A Study of Axicabtagene Ciloleucel and Glofitamab as Second-Line Therapy for Relapsed or Refractory Patients With Large B Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0673; NCI-2024-00209 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — glofitamab; obinutuzumab; axicabtagene ciloleucel; brexucabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axicabtagene Ciloleucel (axi-cel) and Glofitamab (Experimental): Participants will receive glofitamab based on a step-up dosing regimen.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Axi-cel

INTERVENTIONS:
Drug: Glofitamab — Given by IV
  Other Names: RO7082859; RG6026
Drug: Obinutuzumab — Given by IV
  Other Names: GA101; Gazyva; RO5072759
Drug: Axi-cel — Given by IV
  Other Names: Axicabtagene ciloleucel; KTE-C19; KTE-X19

SUMMARY:
To learn if the combination of axicabtagene ciloleucel (axi-cel) and glofitamab as first-line therapy in high-risk LBCL participants or as second-line therapy in LBCL participants can help to control the disease.

DETAILED DESCRIPTION:
Primary Objectives

* To evaluate the safety of axicabtagene ciloleucel (axi-cel) and glofitamab as combination therapy in 2nd line LBCL participants
* To evaluate the effect of axi-cel and glofitamab as combination therapy on the best complete response rate in 2nd line LBCL participants

Secondary Objectives

* To evaluate the effect of axi-cel and glofitamab as combination therapy on overall survival (OS) in 2nd line LBCL participants
* To evaluate the effect of axi-cel and glofitamab as combination therapy on progression free survival in 2nd line LBCL participants
* To evaluate the effect of axi-cel and glofitamab as combination therapy on best overall response rate in 2nd line LBCL participants

Exploratory Objectives

* Characterization of tumors via tumor profiling and antigen density measurement using flow cytometry at baseline
* Characterization of genetic markers via tumor single cell (sc) multiome sequencing and whole exome sequencing (WES) at baseline
* To study the kinetics of circulating tumor DNA (ctDNA) during study progression
* To evaluate the development of anti-axi-cel antibodies during study progression
* To evaluate the effect of glofitamab administration on T cell exhaustion during study progression

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD19- and CD20-positive LBCL, including transformation from indolent lymphomas.
* Have disease that is refractory to or relapsed <=12 months after the completion of first-line chemoimmunotherapy

  • Refractory disease defined as no complete response (CR) to first-line therapy; participants who are intolerant to first-line therapy are excluded
* Progressive disease (PD) as best response to first-line therapy
* Stable disease (SD) as best response after at least 4 cycles of first-line therapy (e.g., 4 cycles of R-CHOP)
* Partial response (PR) as best response after at least 6 cycles, and biopsy-proven residual disease or disease progression ≤ 12 months from completion of therapy

  • Relapsed disease defined as CR to first-line therapy followed by biopsy- proven disease relapse ≤ 12 months of completing first-line therapy.
* Participants must have received first-line therapy including:

  * Anti-CD20 monoclonal antibody
  * An anthracycline containing chemotherapy regimen
* Age 18 or older
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Participants must be willing and able to comply with protocol-mandated hospitalization upon administration of the first dose of glofitamab.
* Adequate bone marrow, renal, hepatic, pulmonary, and cardiac function defined as:

  * Absolute neutrophil count ≥ 1000/μL
  * Platelet count either ≥ 75,000/μL or >50K if documented lymphomatous involvement of bone marrow
  * Absolute lymphocyte count ≥ 100/μL
  * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 30 ml/min
  * Serum alanine aminotransferase and aspartate aminotransferase ≤ 2.5 upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 mg/dL, except in participants with Gilbert's syndrome
  * Cardiac ejection fraction ≥ 45%, no evidence of pericardial effusion (except trace or physiological) as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings
  * No clinically significant pleural effusion
  * Baseline oxygen saturation > 92% on room air
* At least 2 weeks must have elapsed since any prior systemic therapy at the time the participants is planned for leukapheresis.
* Toxicities due to prior therapy must be recovered to Grade 1 or less (except for clinically non-significant toxicities such as alopecia).
* No suspicion of central nervous system (CNS) involvement of lymphoma.
* Participants must be willing and able to comply with protocol-mandated hospitalization upon administration of the first dose of glofitamab and with axi-cel.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with treated secondary CNS lymphoma are eligible if follow-up brain imaging after CNS directed therapy shows no evidence of disease.
* Participants with malignancy ≤2 years, whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Participants should be without any active cardiac symptoms and an ejection fraction >45%, and a clinical risk assessment of cardiac function be class 2B or better using the New York Heart Association Functional Classification.
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
* Participants must agree to either remain completely abstinent or to use two effective contraceptive methods that result in a failure rate of < 1% per year from screening until at least 3 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab (whichever is longer) if the participants is a male. If the participant is a female, effective contraception should be used until at least 18 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab (whichever is longer).
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of cycle-6 (C6) of glofitamab administration, and must refrain from donating sperm during this same period.

  • Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
* Ability to understand and the willingness to sign a written informed consent document.
* Autoimmune disease:

  * Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
  * Participants with a history of disease-related immune thrombocytopenic purpura or autoimmune hemolytic anemia may be eligible for this study.
  * Participants with a history of Type I Diabetes Mellitus who are well controlled (defined as a screening hemoglobin A1c < 8% and no urinary ketoacidosis) are eligible.
  * Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
* Rash must cover < 10% of body surface area
* Disease is well controlled at baseline and requires only low- potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency oral corticosteroids within the previous 12 months
* Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurologic deficits, as judged by the investigator, are allowed

Exclusion Criteria:

* Prior CAR T-cell therapy or glofitamab therapy.
* History of severe, immediate hypersensitivity reaction attributed to aminoglycosides.
* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring hospitalization and/or intravenous (IV) antimicrobials for management within 4 weeks of treatment initiation; simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the sponsor's medical monitor.
* History of uncontrolled human immunodeficiency virus (HIV) infection (HIV+ patients are not excluded from study if they have CD4 counts ≥ 200/µl, are on stable antiretroviral therapy for at least 1 month prior to study entry, and who have an undetectable viral load) or acute or chronic active hepatitis B or C infection; patients with history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America guidelines.
* Presence of any in dwelling line or drain (e.g., percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter); dedicated central venous access catheters, such as a Port-A-Cath® or Hickman® catheter, are permitted.
* Participants with detectable cerebrospinal fluid malignant cells, brain metastases, or active CNS lymphoma.
* History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
* Participants with cardiac lymphoma involvement.
* History of significant or extensive cardiovascular disease such as New York Heart Association Class III or IV cardiac disease or Objective Assessment Class C or D, myocardial infarction within the last 3 months, unstable arrhythmias, or unstable angina.
* Requirement for urgent therapy due to tumor mass effects (e.g., blood vessel compression, bowel obstruction, or transmural gastric involvement).
* Primary immunodeficiency.
* History of autoimmune disease, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment.
* Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to axi-cel, glofitamab, obinutuzumab, or other agents used in the study.
* Administration of a live, attenuated vaccine within 4 weeks before Gpt infusion or anticipation that such a live attenuated vaccine will be required during the study. (Note: Influenza vaccination should be given during influenza season only). Patients must not receive live, attenuated influenza vaccine (e.g., Flumist®) at any time during the study treatment period.
* Participants who have not recovered from AEs due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Participants who are receiving any other investigational agents.
* Women of childbearing potential who are pregnant or breastfeeding. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential.
* Participants who are not willing to practice birth control for the duration of study participation, and 4 months after completion of C6 of glofitamab administration.
* In the investigator's judgment, the participant is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.
* Participants with a known or suspected history of HLH
* Participants with known or suspected chronic active EBV or CMV infection
* Prior treatment with systemic immunotherapeutic agents, including but not limited to radio-immunoconjugates, antibody-drug conjugates, immune/cytokines and monoclonal antibodies (e.g., anti-CTLA4, anti-PD1 and anti-PDL1) within 4 weeks or five half-lives of the drug, whichever is shorter, before Gpt infusion.
* Prior solid organ transplantation
* Participants with history of confirmed progressive multifocal leukoencephalopathy (PML)
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Diagnosis with SARS-CoV-2 infection within 30 days prior to the first study treatment, including asymptomatic SARS-CoV-2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jason Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org